CLINICAL TRIAL: NCT05799976
Title: A Pragmatic Randomized Intervention Using Text Messages Prior to Primary Care Visits to Encourage Care Gap Closure: The PRIME Randomized Clinical Trial
Brief Title: Text Message-Based Nudges Prior to Primary Care Visits to Increase Care Gap Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitesh Patel (Industry)
Responsible Party: Sponsor-Investigator, Mitesh Patel, VP, Ascension, Ascension Health
Organization: Ascension Health (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RIN20230039
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Pneumonia, Pneumococcal; Diabetes Mellitus; Breast Cancer; Colorectal Cancer
MeSH Terms: conditions — Pneumonia, Pneumococcal; Diabetes Mellitus; Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a randomized clinical trial to evaluate a health system initiative to improve care gap closure. We will randomly assign primary care practices that use AthenaClinicals electronic health record at the following locations at Ascension's health system: Alabama-Birmingham, Kansas-Wichita, Tennessee-Nashville, Texas-Austin, and Texas-Waco. These practices will have the opportunity to opt-out from the program before randomization occurs.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): This is a group will serve as usual care and have no intervention during the study period
- Text Message Group (Experimental): This group of primary care practices will be randomized to have the text message intervention
  Interventions: Behavioral: Text message nudge

INTERVENTIONS:
Behavioral: Text message nudge — The text message nudge will be sent to patients 3 days and 1 day prior to a visit with the primary care practices and notify them of up to 3 care gaps based on electronic health record data. Care gaps will be selected based on availability and ranked in this order: influenza vaccination, pneumococcal vaccination, breast cancer screening, colorectal cancer screening, hemoglobin A1 testing, or statin therapy.
  Arms: Text Message Group

SUMMARY:
Primary care visits are a key aspect of clinical care focused on helping patients to close care gaps related to preventive care such as vaccination, diabetes testing, statin therapy and cancer screening. However, less than 50% of care gaps are closed during these visits and new approaches are needed to prime patients for a discussion during these visits. In this study, the study team will evaluate a health system initiative that uses text messaging to patients in days preceding a primary care visit to prime patients to be amenable to ordering of vaccination, diabetes testing, cancer screening, and statin prescribing.

DETAILED DESCRIPTION:
The United States Preventive Services Task Force has recommended tests and treatments for vaccination, diabetes testing, statin therapy, and cancer screening. These preventive services have been demonstrated to reduce illness and improve quality of care. Yet, more than 50% of open care gaps go unaddressed during primary care visits.

Nudges are subtle changes to the way information is framed or choices are offered that can have a significant impact on behavior. In a previous randomized clinical trial, text messages sent to patients prior to primary care visits increased vaccination by up to 11% relative to control. The most effective message told patients the influenza vaccine was "reserved for you," and sent two text messages to patients in the 3 days preceding a primary care appointment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Have documented consent to communicate electronically
* Have a visit scheduled with a primary care practice
* Have at least one open care gap among those in the intervention

Exclusion Criteria:

* No phone number on file to send text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29334 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Care gap order rate | By the end of the day of the primary care visit
  The proportion of open care gaps that have a test or treatment ordered to address them

OTHER OUTCOMES:
Care gap completion rate | Within 3 months of the primary care visit
  The proportion of open care gaps that have a test or treatment completed to address them. Exploratory and only if data is available

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, Principal Investigator — Principal Investigator
Locations (1):
- Ascension, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Has patient information that we are not approved to share

REFERENCES:
- [Background] Milkman KL, Patel MS, Gandhi L, Graci HN, Gromet DM, Ho H, Kay JS, Lee TW, Akinola M, Beshears J, Bogard JE, Buttenheim A, Chabris CF, Chapman GB, Choi JJ, Dai H, Fox CR, Goren A, Hilchey MD, Hmurovic J, John LK, Karlan D, Kim M, Laibson D, Lamberton C, Madrian BC, Meyer MN, Modanu M, Nam J, Rogers T, Rondina R, Saccardo S, Shermohammed M, Soman D, Sparks J, Warren C, Weber M, Berman R, Evans CN, Snider CK, Tsukayama E, Van den Bulte C, Volpp KG, Duckworth AL. A megastudy of text-based nudges encouraging patients to get vaccinated at an upcoming doctor's appointment. Proc Natl Acad Sci U S A. 2021 May 18;118(20):e2101165118. doi: 10.1073/pnas.2101165118. PMID 33926993
- [Derived] Patel MS, Aloia TA, Shoemaker AG, Fakih MG, Masoudi FA, Smith L, Rosenzweig E, Chaiyachati KH, Conrad BN, Bandreddi J, Fogel RI. A Digital Care Plan Nudge to Improve Primary Care Outcomes. NEJM Evid. 2025 Jun;4(6):EVIDoa2400419. doi: 10.1056/EVIDoa2400419. Epub 2025 May 27. PMID 40423396